CLINICAL TRIAL: NCT02977195
Title: NP137 - An Open-label, First in Human, Phase I Trial Aiming to Evaluate the Safety, Pharmacokinetics, and Clinical Activity of a Humanized Monoclonal Antibody Targeting Netrin 1 (NP137) in Patients With Advanced/Metastatic Solid Tumors.
Brief Title: First in Human Evaluation of Safety, Pharmacokinetics, and Clinical Activity of a Monoclonal Antibody Targeting Netrin 1 in Patients With Advanced/Metastatic Solid Tumors
Acronym: NP137
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET15-098 (NP137); 2015-003907-41 (EudraCT Number)
Record Dates: First submitted 2016-11-25; First posted 2016-11-30 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumor; Endometrial Carcinoma; Hormone Receptor Positive
Keywords: First in Human; monoclonal antibody; Netrin-1
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation part, biological cohort and expansion Parts (Experimental): Dose Escalation and Biological Cohort: NP137 was administrated in patients with locally advanced or metastatic solid tumors Expansion Parts: NP137 was administrated in patients with locally advanced or metastatic solid tumors (Expansion part 1) and in patients with RH+ endometrial cancers (Expansion part 2)
  Interventions: Drug: NP137 DL and RP2D

INTERVENTIONS:
Drug: NP137 DL and RP2D — DOSE ESCALATION PART: 7 DL: NP137 was administrated every 2 weeks, as single agent by intravenous injection over 90 min with up to 7 ascending dose levels: Dose level 1: 1 mg/kg Dose level 2: 2 mg/kg Dose level 3: 4 mg/kg Dose level 4: 6 mg/kg Dose level 5: 9 mg/kg Dose level 6: 14 mg/kg Dose level 7: 20 mg/kg
  EXPANSION PARTS: NP137 was administered every 2 weeks, as single agent by intravenous injection over 180 min at 14 mg/kg (RP2D defined in the Dose escalation part).
  FOR ALL PARTS AND COHORT: Treatment will be administered as long as patient experiences clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

SUMMARY:
For most advanced solid tumors, current therapy is inadequate at improving quality of life, slowing progression of disease, prolonging survival, and providing a cure. Hence, there is a continuous need for innovative, safer and more effective anti-cancer therapies. Our study is based on the dependence receptor paradigm and the associated therapeutic strategy. In preclinical models, preventing Netrin-1 interaction with its receptors is sufficient to trigger Netrin-1-expressing tumor cell death in vitro as well as tumor growth and metastasis inhibition in vivo. This indicates that a therapeutic approach based on Netrin-1/Netrin-1 receptors interaction inhibition is both feasible and promising. NP137 is a "first-in-class" humanized monoclonal antibody targeting the Netrin-1 ligand, a secreted protein recently described as a driver of tumor initiation and progression. NP137 demonstrated anti-tumor activity as a single agent in several pre-clinical models of cancer, including breast and lung cancer. Taken together, several studies strongly support the rational for preclinical development and clinical evaluation of a highly potent and selective anti-Netrin-1 antibody in cancer patients. The proposed study is an open label, multicenter, Phase I dose escalation study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) and preliminary anti-tumor activity of NP137 administered every 2 weeks (Q2W) as single agent in patients with locally advanced or metastatic solid tumors. This trial will be the First in Human (FIH) study for NP137; there is no clinical experience with this antibody in the clinic. The study consists of 3 parts:

Part 1) a dose escalation part to define the Maximum tolerated dose and the Recommended Phase II dose (MTD /RP2D) of NP137 as well as to research some PD biomarkers (Biological collection cohorts) - This part is now completed with Last Patient In on December 20th 2018 - Part 2) an expansion part#1 to investigate NP137 clinical activity as a single agent by collecting the 3-month objective response rate (ORR3m).

Part 3) an expansion part#2 to investigate NP137 clinical activity as a single agent by collecting the 3-month objective response rate (ORR3m) in RH+ patients with endometrial carcinoma.

DETAILED DESCRIPTION:
The dose escalation part (NP137 administered as a single agent by intravenous injection with 7 ascending dose levels) has been initiated with an accelerated dose titration with 1 patient per DL until the occurrence of a ≥ Grade 2 drug-related AE. Following the occurrence of such moderate toxicity, patients have been enrolled in a slower dose escalation design with at least 3 patients per DL using a Modified Continual Reassessment Method. Of note, in case no toxicity occurs up to the DL4, the classical 3+3 design has been initiated. Cohorts of patients with biopsable disease have been added in order to assess the impact of NP137 treatment on epithelial phenotype signature (assessed by RNAseq and subsequent bioinformatic profiling using published E vs M score). Up to 4 additional and independent cohorts of patients (n= up to 6 pts/ cohort) with biopsable disease have been enrolled. Starting from DL4, the enrolment in such cohort will be allowed at highest DL that has cleared its DLT assessment window. Such cohorts will allow to collect pre and on-treatment tumor biopsies in order to identify PD biomarkers correlated to NP137 clinical activity.

In expansion parts, patients are treated at the RP2D defined in Part 1 (14 mg/kg).

In both parts, NP137 will continue to be administered as long as patient experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent or patient willingness to stop the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥ 18 years at time of inform consent signature.
* For dose escalation cohorts, biological cohorts ans extension parts: Histological confirmed locally advanced/metastatic solid tumors of any histological types.

For second expansion part only: patients with histologically confirmed locally advanced / metastatic endometrial carcinoma and who positively expressed Hormone Receptors (with a positivity threshold value ≥ 10%). Estrogene receptors (ER) and Progesterone Receptors (PR) expression rates must be assessed by immunohistochemistry and fully documented.

* Documented disease progression after at least one prior line of treatment in the metastatic/advanced setting.
* Patient must be, in the judgment of the investigator, an appropriate candidate for an experimental therapy i.e. with no available curative options.
* At least one measurable lesion as per RECIST 1.1.
* For Expansion part only: Availability of at least 2 pre-treatment scans prior to C1D1 including the screening scan (i.e. within 28 days before C1D1) and the most recent scan prior to screening to evaluate tumor growth kinetics.
* Mandatory for Biological collection cohorts and Expansion part #1 and #2 only (optional for dose escalation): Availability of a representative archival tumor specimen in formalin-fixed paraffin embedded (FFPE) block with an associated pathology report. Optional for Expansion part #2 only (RH+ endometrial carcinoma] Biopsable disease i.e. at least one lesion with a diameter ≥10 mm, visible by medical imaging and accessible to percutaneous sampling.
* Life expectancy ≥ 12 weeks.
* ECOG PS 0-1
* Adequate hematological function: Hemoglobin ≥ 9 g/dL, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelet count ≥ 100 x 109/L (without transfusion within 21 days before C1D1).
* Adequate renal function: Calculated creatinine clearance by MDRD or CDK-EPI ≥50 mL/min/1.73m2 or serum creatinine ≤ 1.5 ULN
* Adequate liver function: AST and ALT ≤ 2.5 ULN (up to 5 ULN may be tolerated in case of liver metastases), Total serum bilirubin ≤ 1.5 x ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤3mg/dL is acceptable).
* Adequate coagulation function: INR≤ 1.5, aPTT≤ 1.5 ULN.
* Adequate cardiovascular function: QTc ≤470ms, Resting BP systolic <160mmHg and diastolic<100mmHg, LVEF ≥50% as determined by multiple-gated acquisition (MUGA) scan or transthoracic echocardiogram
* Minimal wash-out period for prior treatment before C1D1: For chemotherapy, tyrosine kinase inhibitor > 2 weeks, Radiation therapy >4 weeks, For monoclonal antibodies >4 weeks, For immunosuppressive medication > 2 weeks, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at doses which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, Major surgery >4 weeks, For hormonotherapy > 2 weeks with exception of GnRH analogs for prostate cancer patients who should continue on GnRH analogs throughout the study.
* Women of child-bearing potential must have a negative serum pregnancy test at screening (7 days before C1D1).
* Women of child-bearing potential must agree to remain abstinent or to use 2 effective forms of contraception from the time of the negative pregnancy test up to 3 months after the last dose of study drug. Effective forms of contraception are listed in Protocol.
* Men must agree to remain abstinent or to use an effective contraceptive method during the study and for up to 3 months after the last dose of study drug
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures.
* Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Persistence of CTCAE ≥ Grade 2 toxicity due to prior anti-cancer therapy (except alopecia (any grades), blood tests values according to inclusion criteria, Grade ≥3 peripheral neuropathy.
* History of severe allergic anaphylactic reactions to one of the components of the study drug or to humanized mAbs
* Any known neurodegenerative (Alzheimer's disease, Parkinson's disease and related disorders, amyotrophic lateral sclerosis, prion disease, motor neuron diseases, Huntington's disease, spinocerebellar ataxia, spinal muscular atrophy,) or neuroinflammatory disease (multiple sclerosis, …).
* Active or untreated CNS metastases. Patients with radiographically stable, asymptomatic previously irradiated lesions are eligible provided that patient is ≥ 4 weeks beyond completion of cranial irradiation and ≥ 3 weeks off of corticosteroid therapy are eligible.
* Any uncontrolled intercurrent illness that would limit compliance with protocol requirements including, but not limited to: Ongoing or active infection including acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), History of chronic liver disease or hepatic cirrhosis, Impaired cardiovascular function or clinically significant cardiovascular diseases including but not limited to symptomatic congestive heart failure, history of acute myocardial infection, acute coronary syndromes; history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality within 6 months prior to C1D1, Psychiatric illness / specific social situations.
* Other invasive malignancy in the last 2 years except for those with a minimal risk of metastasis or death such as adequately managed in-situ carcinoma of the cervix, basal or squamous cell skin cancer, localized prostate cancer or ductal carcinoma in situ treated with curative intent.
* Needs to be treated with a forbidden concomitant/concurrent therapies/procedures including: Any investigational anticancer therapy other than the study drug , Any concurrent chemotherapy, radiotherapy (except palliative radiotherapy performed on non-target lesion and following sponsor's approval), immunotherapy, biologic or hormonal therapy* for cancer treatment. *: for prostate cancer patients, treatment with GnrH analogs is allowed, Immunosuppressive medications including methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications including steroids for the management of AEs or in subjects with contrast allergies is acceptable, Major surgery, Any hematopoietic growth factor (during the DLT period)
* Female subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Part 1 (dose escalation part): DLT occurrence | At the end of Cycle 2 (each cycle is 14 days)
  Dose Limiting toxicities (DLTs) are any pre-defined toxicities graded by using NCI-CTCAE v4.0 occurring during the DLT period (i.e . 28 days) and assessed as related to study drug and any other study drug related toxicity considered significant enough to be qualified as DLT in the opinion of the investigators after discussion with the sponsor. Indeed, as a principle in this first in Man study, any toxicity that the investigator or the sponsor determines to be dose-limiting, regardless of the grade, may be considered as a DLT.
Part 2 (expansion part #1): Objective response rate after 3 months | 12 weeks of treatment (=3 months)
  Objective response rate after 3 months (ORR3m) is defined as the rate of patients with complete response (CR) or partial response (PR) after 3 months of treatment (measurements according to RECIST 1.1 criteria).
Part 3 (expansion part #2): Objective response rate after 3 months in RH+ patients with endometrial carcinoma | 12 weeks of treatment (=3 months)
  Objective response rate after 3 months (ORR3m) is defined as the rate of patients with complete response (CR) or partial response (PR) after 3 months of treatment (measurements according to RECIST 1.1 criteria).

SECONDARY OUTCOMES:
Adverse events reporting | from the date of first intake of study drug until 90 days after study drug discontinuation or at time of initiation of a new anti-cancer treatment
  Any adverse events (AEs) graded according to NCI-CTCAE, Version 4.03.
Overall response Rate (ORR) | from the date of first study drug intake until until first documented progression, assessed up to 52 weeks
  Overall response Rate (ORR) is the proportion of evaluable patients with objective response i.e. CR or PR according to RECIST 1.1.
Duration of Response (DoR) | from the time of first objective response (CR or PR as per RECIST 1.1 criteria) until first documented progression, assessed up to 52 weeks
  Time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression or death is documented,
Clinical Benefit Rate (CBR) | from the date of first study drug intake until until first documented progression, assessed up to 52 weeks
  Clinical Benefit Rate (CBR) is the proportion of evaluable patients with an objective response i.e. CR, PR or SD according to RECIST 1.1.
Progression-free survival (for expansion part only) | from the date of first study drug intake until disease progression or death, whichever occurs first, up to 52 weeks
  Time from first study drug intake until disease progression or death, whichever occurs first
PFS2/PFS1 (for expansion part only) | From the date of first intake of previous treatment before inclusion until disease progression or death, whichever occurs first, up to 52 weeks
  PFS2/PFS1 is defined as the ratio of the PFS of the current treatment (PFS2) versus the PFS of previous treatment before inclusion (PFS1).
Tumor Growth Kinetics (growth rate) | from date of progression under previous treatment before inclusion until disease progression, up to 52 weeks
  An exploratory assessment of tumor growth kinetics will be made by comparing post-treatment scans with at least 2 pre-treatment scans.
Area under the NP137 plasma concentration (AUC) versus time curve | Over the first 6 cycles (each cycle is 14 days) and 30 days after last study drug intake
  Area under the concentration-time curve from time zero to the last sample with the quantifiable concentration.
Peak NP137 plasma concentration (Cmax) | Over the first 6 cycles (each cycle is 14 days) and 30 days after last study drug intake
  Plasma peak concentration of NP137
NP137 terminal elimination half-time (t1/2) | Over the first 6 cycles (each cycle is 14 days) and 30 days after last study drug intake
  Terminal elimination half-life: time required for the amount of NP137 in the body to decrease by half.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Ico - Rene Gauducheau, Nantes
  - IUCT-Oncopôle de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lengrand J, Pastushenko I, Vanuytven S, Song Y, Venet D, Sarate RM, Bellina M, Moers V, Boinet A, Sifrim A, Rama N, Ducarouge B, Van Herck J, Dubois C, Scozzaro S, Lemaire S, Gieskes S, Bonni S, Collin A, Braissand N, Allard J, Zindy E, Decaestecker C, Sotiriou C, Salmon I, Mehlen P, Voet T, Bernet A, Blanpain C. Pharmacological targeting of netrin-1 inhibits EMT in cancer. Nature. 2023 Aug;620(7973):402-408. doi: 10.1038/s41586-023-06372-2. Epub 2023 Aug 2. PMID 37532929
- [Derived] Sun Y, Manceau A, Frydman L, Cappuccio L, Neves D, Basso V, Wang H, Fombonne J, Maisse C, Mehlen P, Paradisi A. Delta40p53 isoform up-regulates netrin-1/UNC5B expression and potentiates netrin-1 pro-oncogenic activity. Proc Natl Acad Sci U S A. 2021 Sep 7;118(36):e2103319118. doi: 10.1073/pnas.2103319118. PMID 34470826